CLINICAL TRIAL: NCT00750009
Title: Preparatory Aid to Improve Decision Making About Cancer Clinical Trials (PRE-ACT)
Brief Title: Personalized Information or Basic Information in Helping Patients Make Decisions About Participating in a Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CASE18Z09; R01CA127655 (NIH); FCCC-08808 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Brain and Central Nervous System Tumors; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage 0 chronic lymphocytic leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated hairy cell leukemia; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage II childhood lymphoblastic lymphoma; stage II childhood small noncleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III childhood large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; Burkitt lymphoma; childhood diffuse large cell lymphoma; childhood grade III lymphomatoid granulomatosis; childhood immunoblastic large cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; childhood myelodysplastic syndromes; recurrent childhood anaplastic large cell lymphoma; stage I childhood anaplastic large cell lymphoma; stage II childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Recurrence; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Dendritic Cell Sarcoma, Interdigitating; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Immunoglobulin Light-chain Amyloidosis | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (PRE-ACT) (Experimental): Patients receive tailored feedback and video content to address clinical trial barriers following baseline assessment.
  Interventions: Other: educational intervention
- Arm II (control) (Active Comparator): Patients receive generic clinical trials educational feedback taken from NCI publications following baseline assessment.
  Interventions: Other: educational intervention

INTERVENTIONS:
Other: educational intervention — Patients receive a tailored intervention or generic information

SUMMARY:
RATIONALE: Providing information that is tailored to answer patients' questions about clinical trials may help patients with cancer decide to enroll in a clinical trial. It is not known whether providing personalized information is more effective than basic information in helping patients make decisions about clinical trials.

PURPOSE: This randomized phase III trial is studying personalized information to see how well it works compared with basic information in helping patients make decisions about participating in a clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To improve preparation for consideration of clinical trials by providing tailored information to address barriers related to knowledge, goals and values, and beliefs and expectancies before their physician visit in patients with advanced metastatic or early stage cancer.

Secondary

* To develop and pilot test a tailored interactive preparatory aid (PRE-ACT) to promote informed cancer treatment decision making by addressing barriers to considering clinical trials as a treatment option.
* To evaluate the efficacy of PRE-ACT in improving preparation for considering participation in clinical trials by conducting a randomized clinical trial to compare PRE-ACT vs generic clinical trial information with text (control condition).
* To investigate relevant background and psychosocial variables that are associated with preparedness, barriers, and treatment outcomes.
* To investigate the impact of PRE-ACT on patient decisional conflict, satisfaction with information received, satisfaction with discussion about clinical trials with the physician, satisfaction with the treatment decision, clinical trials discussion, clinical trials participation, and quality of informed consent.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (PRE-ACT): Patients receive tailored feedback and video content to address clinical trial barriers following baseline assessment.
* Arm II (control): Patients receive generic clinical trials educational feedback taken from NCI publications following baseline assessment.

All patients complete a baseline assessment to assess demographics, personal characteristics, preparedness, and barriers to clinical trials. All patients also undergo a post-intervention assessment and complete a survey to measure preparedness for consideration of clinical trials, and impact of the intervention on clinical trials barriers. A brief patient post-consultation assessment is completed by patients within two weeks of the physician consultation to determine whether clinical trials were discussed, patient satisfaction with discussion about clinical trials, treatment options, treatment selection, decisional conflict, and satisfaction with treatment decision. Quality of informed consent is also assessed for patients participating in a clinical trial and completing the consent process during their initial physician consultation. Each patient's physician completes a brief Physician Post-Consultation Assessment to define cancer stage, treatment goal, and to determine whether clinical trials were offered and accepted and if not, why not. For patients who have not made a treatment decision after consultation, a brief follow-up phone survey or medical chart review is used to identify the patient's treatment choice.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Advanced (metastatic) disease
  * Early stage (i.e., appropriate for adjuvant therapy) disease
* Scheduled for first outpatient consultation with a medical oncologist at the Clinical Centers

PATIENT CHARACTERISTICS:

* Able to read and verbally communicate in English
* Patients who choose to complete the intervention at home rather than at the Clinical Center before their visit must have high-speed (i.e., DSL or cable) Internet access

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement in preparation for consideration of clinical trials | after pts.complete all survey measures

SECONDARY OUTCOMES:
Development and pilot testing of a tailored interactive preparatory aid (PRE-ACT) | after pts.complete all survey measures
Efficacy of PRE-ACT | after pts.complete all survey measures
Comparison of PRE-ACT and genomic clinical trial information with text | after pts.complete all survey measures
Relevant background and psychosocial variables that are associated with preparedness, barriers, and treatment outcomes | after pts.complete all survey measures
Impact of PRE-ACT on patient | after pts.complete all survey measures
  To investigate the impact of PRE-ACT on patient decisional conflict, satisfaction with information received, satisfaction with discussion about clinical trials with the physician, satisfaction with the treatment decision, clinical trials discussion, clinical trials participation, and quality of informed consent. (Exploratory Aim)

CONTACTS AND LOCATIONS:
Overall Officials: Neal J. Meropol, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Meropol NJ, Wong YN, Albrecht T, Manne S, Miller SM, Flamm AL, Benson AB 3rd, Buzaglo J, Collins M, Egleston B, Fleisher L, Katz M, Kinzy TG, Liu TM, Margevicius S, Miller DM, Poole D, Roach N, Ross E, Schluchter MD. Randomized Trial of a Web-Based Intervention to Address Barriers to Clinical Trials. J Clin Oncol. 2016 Feb 10;34(5):469-78. doi: 10.1200/JCO.2015.63.2257. Epub 2015 Dec 23. PMID 26700123
- [Derived] Wong YN, Schluchter MD, Albrecht TL, Benson AB 3rd, Buzaglo J, Collins M, Flamm AL, Fleisher L, Katz M, Kinzy TG, Liu TM, Manne S, Margevicius S, Miller DM, Miller SM, Poole D, Raivitch S, Roach N, Ross E, Meropol NJ. Financial Concerns About Participation in Clinical Trials Among Patients With Cancer. J Clin Oncol. 2016 Feb 10;34(5):479-87. doi: 10.1200/JCO.2015.63.2463. Epub 2015 Dec 23. PMID 26700120